CLINICAL TRIAL: NCT05588128
Title: A Study of Prospective Monitoring of Subjects With Biochemically Recurrent Prostate Cancer Using 18F-DCFPyL
Brief Title: Prospective Monitoring of Subjects With Biochemically Recurrent Prostate Cancer Using 18FDCFPyL
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000628; 000628-C
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Prostate Cancer; Biochemically Recurrent
Keywords: Cancer Of Prostate; Natural History; Imaging
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with biochemically recurrent prostate cancer
  Interventions: Drug: 18F-DCFpyL

INTERVENTIONS:
Drug: 18F-DCFpyL — Administered to Cohort.

SUMMARY:
Background:

Prostate cancer is the second leading cause of cancer-related death in American men. The disease recurs in up to 50,000 men each year after their early-stage disease was treated; however, at this stage, imaging scans are often unable to find the disease in the body. In this natural history study, researchers want to find out if a new radiotracer (18F-DCFPyL) injected before positron emission tomography (PET) imaging can help identify sites in the body with cancer.

Objective:

To learn more about how 18F-DCFPyL PET/CT scans detect change over time in men with recurrent prostate cancer.

Eligibility:

Men aged 18 and older with prostate cancer that returned after treatment.

Design:

Participants will be screened with blood tests. They will also have a bone scan and a computed tomography (CT) scans of the chest, abdomen, and pelvis.

Participants will have an initial study visit. They will have a physical exam and blood tests. They will have a PET/CT scan with 18F-DCFPyL. The radiotracer will be injected into a vein; this will take about 20 seconds. The PET/CT scan will be done 1 to 2 hours later. Participants will lie still on a scanner table while a machine captures images of their body. The scan will take 45 minutes.

Participants will return for blood tests every 3 months.

Participants will return for additional scans with 18F-DCFPyL on this schedule:

Once a year if their previous scan was negative for prostate cancer.

Every 6 months if their previous scan was positive for prostate cancer.

Participants may be in the study up to 5 years.

DETAILED DESCRIPTION:
Background:

* Prostate cancer is the most common malignancy and the second leading cause of cancer-related deaths in American men.
* About 25,000 to 50,000 men each year develop a rising prostate-specific antigen (PSA) after definitive radiation or surgery for early-stage disease but have negative findings on computed tomography (CT) and Tc99 bone scan (standard imaging in prostate cancer).
* The recent Food and Drug Administration (FDA) approval of 18F-DCFPyL PET imaging provides an opportunity to locate micrometastatic lesions in patients with recurrent disease.
* It is unknown how these lesions (or prostate cancer) evolve over time in men with positive findings on 18F-DCFPyL PET imaging.

Objective:

-To observe participants with biochemically recurrent prostate cancer for 5 years to understand the evolution of 18F-DCFPyL PET lesions in this population.

Eligibility:

* History of primary treatment for prostate cancer (either surgery or radiation).
* PSA >= 0.50, and testosterone >100.
* Age >=18 years.
* No evidence of metastatic soft tissue disease on CT scan (or MRI), or bone lesions on bone scan.
* No androgen deprivation therapy (ADT), no systemic therapy within the 6 months before the study intervention, and no prostatectomy within 1 year before the study intervention.

Design:

* Eligible participants will have clinical evaluations and imaging studies. Participants with negative findings on initial/following 18F-DCFPyL scan(s) will be invited approximately every year (+/-12 weeks) for follow-up imaging studies (including 18F-DCFPyL PET scans). Participants with positive findings on initial/following 18F-DCFPyL scan(s) will be invited approximately every 6 months (+/-8 weeks) for repeat scans, not to exceed 2 scans per year.
* After the initial evaluation, participants will be invited to NIH approximately every 3 months (+/- 4 weeks) for PSA testing.

ELIGIBILITY:
* INCLUSION CRITERIA:
* History of primary treatment for prostate cancer (either surgery or radiation)
* Serum PSA >= 0.50
* Serum testosterone >100
* Age >=18 years
* Men must agree to use highly effective contraception (surgical sterilization) for 7 days after every study agent administration. Note: abstinence, defined as no heterosexual sexual intercourse when this is in line with the preferred and usual lifestyle of the subject is also acceptable
* The ability of a participant to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

-Evidence of soft tissue disease on CT scan (or magnetic resonance imaging [MRI] as clinically indicated).

NOTE: Lymph nodes <= 1.5 cm in the shortest dimension are allowed.

* Evidence of bone lesions on Tc99 bone scan
* Prostatectomy within 1 year before the study intervention
* Androgen deprivation therapy (ADT) within the 6 months before the study intervention
* Systemic therapy for prostate cancer within the 6 months before the study intervention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Observation of 18F-DCFPyL lesions in BRPC | baseline through 5 years
  Initial 18F-DCFPyL imaging, every 6 months (+/- 8 weeks) for participants positive on imaging, and every 12 months (+/- 12 weeks) for participants negative on imaging until 5 years.

SECONDARY OUTCOMES:
Progression on 18F-DCFPyL | baseline through 5 years
  Initial 18F-DCFPyL imaging, every 6 months (+/- 8 weeks) for participants positive on imaging, and every 12 months (+/- 12 weeks) for participants negative on imaging until 5 years.
Evaluate PSA doubling in association with 18F-DCFPyL changes | baseline through 5 years
  PSA test every 3 months (+/- 4 weeks) until 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing will be shared with subscribers to dbGAP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be made available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000628-C.html